CLINICAL TRIAL: NCT03762850
Title: A Randomized, Multicenter, Double-blind, Parallel-group, Active-control Study of the Efficacy and Safety of Sparsentan for the Treatment of Immunoglobulin A Nephropathy
Brief Title: A Study of the Effect and Safety of Sparsentan in the Treatment of Patients With IgA Nephropathy
Acronym: PROTECT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Travere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 021IGAN17001; 2017-004605-41 (EudraCT Number)
Record Dates: First submitted 2018-11-27; First posted 2018-12-04 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Immunoglobulin A Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — sparsentan; Irbesartan; dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- sparsentan (Experimental): Double-blind: Sparsentan will be administered daily as a 200-mg oral tablet, over-encapsulated (blinded) size 00 capsule for the first 2 weeks of the study following randomization. For patients who tolerate the initial dose of 200 mg after 2 weeks will increase their dose to 400- mg and continue treatment to Week 110.
  Interventions: Drug: sparsentan
- irbesartan (Active Comparator): Double-blind: Irbesartan will be administered daily as a 150-mg oral tablet, over-encapsulated (blinded) size 00 capsule for the first 2 weeks of the study following randomization. For patients who tolerate the initial dose of 150 mg after 2 weeks will increase their dose to 300 mg and continue treatment to Week 110.
  Interventions: Drug: irbesartan
- dapagliflozin + sparsentan (Sub study) (Experimental): OLE Sub study: Dapagliflozin will be administered daily as a 5-mg oral tablet, in addition to 400-mg of Sparsentan, for a period of 12 weeks.
  Interventions: Drug: sparsentan; Drug: Dapagliflozin
- sparsentan (Sub Study) (Experimental): OLE Sub study: Sparsentan will be administered daily as a dose of 400-mg for a period of 12 weeks.
  Interventions: Drug: sparsentan

INTERVENTIONS:
Drug: sparsentan — Target dose of 400 mg daily
  Other Names: RE-021
  Arms: dapagliflozin + sparsentan (Sub study); sparsentan; sparsentan (Sub Study)
Drug: irbesartan — Target dose of 300 mg daily
  Other Names: Irbesartan Tablets USP
  Arms: irbesartan
Drug: Dapagliflozin — Target dose of 10 mg daily
  Arms: dapagliflozin + sparsentan (Sub study)

SUMMARY:
To determine the long-term (approximately 2 years) nephroprotective potential of treatment with sparsentan as compared to an angiotensin receptor blocker in patients with immunoglobulin A nephropathy (IgAN).

DETAILED DESCRIPTION:
This is a 114-week,randomized, multicenter, double-blind, parallel-group, active-control study with an open-label extension period of up to 156 weeks, for a total duration of up to 270 weeks in patients with IgAN who have persistent overt proteinuria and remain at high risk of disease progression despite being on a stable dose (or doses) of an angiotensin-converting enzyme inhibitor (ACEI) and/or angiotensin receptor blocker (ARB) that is (are) a maximum tolerated dose that is at least one half of the maximum labeled dose (MLD) (according to approved labeling. Approximately 380 patients aged ≥18 years will be enrolled in the study globally. The investigational drug (sparsentan) is a dual acting angiotensin receptor blocker and endothelin receptor antagonist. The active control is irbesartan.

The purpose of the study is to evaluate the potential benefit of sparsentan on kidney function by analyzing change in proteinuria (protein in urine) and estimated glomerular filtration rate (eGFR) as compared to current standard treatment.

Patients enrolled in the PROTECT study (Protocol 021IGAN17001) will be those at high risk of progressing to renal failure. They will be randomly assigned in a 1:1 ratio to either sparsentan or irbesartan, as the active control (current standard treatment) at the Day 1 (Randomization) visit. Study medication (sparsentan and irbesartan) will be administered as a single oral morning dose.

The primary analysis is change in proteinuria (urine protein/creatinine ratio) from baseline at Week 36 in sparsentan-treated patients as compared to irbesartan-treated patients.

Primary completion date represents the anticipated completion date of the double-blind portion of the study. Study completion date represents the anticipated completion date of the open-label extension portion of the study.

Patients participating in the open-label extension period may be evaluated for eligibility to participate in a randomized, open-label, controlled Sub study evaluating the safety and efficacy of an SGLT2 inhibitor in addition to stable sparsentan treatment (OLE Sub study). The SGLT2 inhibitor, dapagliflozin will be provided as "study medication" for the OLE Sub study. Following completion of the visit 12 weeks after the OLE baseline visit, eligible patients may receive open-label dapagliflozin for at least 12 weeks but up to 24 additional weeks, or through the end of the open-label extension period, whichever is shortest. Approximately 60 patients from the open-label extension period will be enrolled into the OLE Sub study.

ELIGIBILITY:
Key Inclusion Criteria for the Double-Blind Period:

* Age 18 years or older at screening
* Biopsy-proven primary IgAN
* Proteinuria of ≥1 g/day at screening
* eGFR ≥30 mL/min/1.73 m2 at screening
* Currently on stable dose of ACEI and/or ARB therapy, for at least 12 weeks prior to screening (maximum tolerated dose and at least one-half of the maximum labeled dose)
* Systolic BP ≤150 mmHg and diastolic BP ≤100 mmHg at screening
* Willing to undergo change in ACEI and/or ARB and anti-hypertensive medications
* Agree to contraception

Key Exclusion Criteria for the Double-Blind Period:

* IgAN secondary to another condition
* Presence of cellular glomerular crescents in >25% of glomeruli on renal biopsy (if biopsy available within 6 months of screening)
* Chronic kidney disease (CKD) in addition to IgAN
* History of organ transplantation, with exception of corneal transplants
* Require any prohibited medications
* Treatment of systemic immunosuppressive medications (including corticosteroids) for >2 weeks within 3 months of screening
* History of heart failure or previous hospitalization for heart failure or unexplained dyspnea, orthopnea, paroxysmal nocturnal dyspnea, ascites, and/or peripheral edema
* Clinically significant cerebrovascular disease or coronary artery disease within 6 months of screening
* Jaundice, hepatitis, or known hepatobiliary disease or elevations of transaminases (ALT/AST) >2 times upper limit of normal at screening
* History of malignancy other than adequately treated basal cell or squamous cell skin cancer or cervical carcinoma within the past 2 years
* Hematocrit value <27% (0.27 V/V) or hemoglobin value <9 g/dL (90 g/L) at Screening
* Potassium >5.5 mEq/L (5.5 mmol/L) at Screening
* History of alcohol of illicit drug use disorder
* History of serious side effect or allergic response to any angiotensin II antagonist or endothelin receptor antagonist, including sparsentan or irbesartan, or has a hypersensitivity to any of the excipients in the study medications
* For female: Pregnancy, or planning to become pregnant during the course of the study, or breastfeeding
* Participation in a study of another investigational product within 28 days of screening

Key Inclusion Criteria for the Open-Label Extension Period based on assessments at the Week 110 visit:

* Completed participation in the double-blind period, including the Week 114 visit
* Did not permanently discontinue study medication during the double-blind period
* Agree to contraception

Key Exclusion Criteria for the Open-Label Extension Period based on assessments at the Week 110 and Week 114 visits:

* Progression to end-stage renal disease (ESRD) requiring renal replacement therapy (RRT)
* Development of any criteria for discontinuation of study medication or discontinuation from the study, between Week 110 and Week 114
* Patient was unable to initiate, or developed contraindications to, treatment with RAAS inhibitors between Week 110 and Week 114
* eGFR ≤20 mL/min/1.73 m2 at Week 110
* Female patient is pregnant or breastfeeding

Key Inclusion Criteria for the OLE Sparsentan + SGLT2 Inhibitor Sub study:

* Participating in the open-label extension and is willing and able to provide signed informed consent for participation in the open-label extension period Sub study
* A urine protein excretion value of ≥0.3 g/day.
* An eGFR of ≥25 mL/min/1.73m2
* On a stable dose of sparsentan for ≥8 weeks in the open-label extension period that is the maximum tolerated dose.

Key Exclusion Criteria for the OLE Sparsentan + SGLT2 Inhibitor Sub study:

* Progressed to ESRD requiring RRT
* Initiated or changed dose of a systemic immunosuppressive medication (including systemic steroids) within 12 weeks
* Taking an SGLT2 inhibitor within 12 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2018-12-11 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2026-07 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Radko Komers, MD, PhD, Study Director — Travere Therapeutics, Inc.
Locations (140):
- United States (37):
  - Travere Investigational Site, Birmingham, Alabama
  - Travere Investigational Site, Homewood, Alabama
  - Travere Investigational Site, Glendale, California
  - Travere Investigational Site, Montebello, California
  - Travere Investigational Site, Northridge, California
  - Travere Investigational Site, San Diego, California
  - Travere Investigational Site, Stanford, California
  - Travere Investigational Site, Denver, Colorado
  - Travere Investigational Site, Coral Springs, Florida
  - Travere Investigational Site, Hollywood, Florida
  - Travere Investigational Site, Miami, Florida
  - Travere Investigational Site, Winter Park, Florida
  - Travere Investigational Site, Lawrenceville, Georgia
  - Travere Investigational Site, Nampa, Idaho
  - Travere Investigational Site, Hinsdale, Illinois
  - Travere Investigational Site, Muncie, Indiana
  - Travere Investigational Site, Kansas City, Kansas
  - Travere Investigational Site, Louisville, Kentucky
  - Travere Investigational Site, Boston, Massachusetts
  - Travere Investigational Site, Springfield, Massachusetts
  - Travere Investigational Site, Worcester, Massachusetts
  - Travere Investigational Site, Minneapolis, Minnesota
  - Travere Investigational Site, Reno, Nevada
  - Travere Investigational Site, Fresh Meadows, New York
  - Travere Investigational Site, New York, New York
  - Travere Investigational Site, Cleveland, Ohio
  - Travere Investigational Site, Columbus, Ohio
  - Travere Investigational Site, Philadelphia, Pennsylvania
  - Travere Investigational Site, Columbia, South Carolina
  - Travere Investigational Site, El Paso, Texas
  - Travere Investigational Site, Fort Worth, Texas
  - Travere Investigational Site, Houston, Texas
  - Travere Investigational Site, Lewisville, Texas
  - Travere Investigational Site, San Antonio, Texas
  - Travere Investigational Site, Salt Lake City, Utah
  - Travere Investigational Site, Tacoma, Washington
  - Travere Investigational Site, Marshfield, Wisconsin
- Australia (10):
  - Travere Investigational Site, Concord, New South Wales
  - Travere Investigational Site, Gosford, New South Wales
  - Travere Investigational Site, Kingswood, New South Wales
  - Travere Investigational Site, New Lambton Heights, New South Wales
  - Travere Investigational Site, Randwick, New South Wales
  - Travere Investigational Site, St Leonards, New South Wales
  - Travere Investigational Site, Birtinya, Queensland
  - Travere Investigational Site, Adelaide, South Australia
  - Travere Investigational Site, Reservoir, Victoria
  - Travere Investigational Site, Nedlands, Western Australia
- Belgium (6):
  - Travere Investigational Site, Bonheiden
  - Travere Investigational Site, Bruges
  - Travere Investigational Site, Ghent
  - Travere Investigational Site, Kortrijk
  - Travere Investigational Site, Liège
  - Travere Investigational Site, Roeselare
- Croatia (2):
  - Travere Investigational Site, Osijek
  - Travere Investigational Site, Zagreb
- Travere Investigational Site, Prague, Czechia
- Estonia (2):
  - Travere Investigational Site, Tallinn
  - Travere Investigational Site, Tartu
- France (8):
  - Travere Investigational Site, Marseille, Bouches-du-Rhone
  - Travere Investigational Site, Montpellier, Herault
  - Travere Investigational Site, Grenoble, Isere
  - Travere Investigational Site, Paris, Paris
  - Travere Investigational Site, Saint-Priest-en-Jarez, Pays de la Loire Region
  - Travere Investigational Site, Clermont-Ferrand, Puy De Dome
  - Travere Investigational Site, Créteil
  - Travere Investigational Site, Paris
- Germany (9):
  - Travere Investigational Site, Villingen-Schwenningen, Baden-Wurttemberg
  - Travere Investigational Site, Hanover, Lower Saxony
  - Travere Investigational Site, Aachen, North Rhine-Westphalia
  - Travere Investigational Site, Düsseldorf, North Rhine-Westphalia
  - Travere Investigational Site, Kaiserslautern, Rheinland Palatinate
  - Travere Investigational Site, Trier, Rheinland Palatinate
  - Travere Investigational Site, Kiel, Schleswig-Holstein
  - Travere Investigational Site, Jena, Thuringia
  - Travere Investigational Site, Berlin
- Hong Kong (5):
  - Travere Investigational Site, Kwun Tong, Kowloon
  - Travere Investigational Site, Lai Chi Kok, Kowloon
  - Travere Investigational Site, Shatin, New Territories
  - Travere Investigational Site, Tsuen Wan, New Territories
  - Travere Investigational Site, Hong Kong
- Italy (10):
  - Travere Investigational Site, Ranica, Bergamo
  - Travere Investigational Site, Milan, Lombardy
  - Travere Investigational Site, Bari
  - Travere Investigational Site, Catania
  - Travere Investigational Site, Catanzaro
  - Travere Investigational Site, Lecco
  - Travere Investigational Site, Modena
  - Travere Investigational Site, Pavia
  - Travere Investigational Site, Roma
  - Travere Investigational Site, Torino
- Lithuania (2):
  - Travere Investigational Site, Kaunas
  - Travere Investigational Site, Vilnius
- New Zealand (4):
  - Travere Investigational Site, Grafton, Auckland
  - Travere Investigational Site, Hamilton
  - Travere Investigational Site, Hastings
  - Travere Investigational Site, New Plymouth
- Poland (5):
  - Travere Investigational Site, Krakow
  - Travere Investigational Site, Lodz
  - Travere Investigational Site, Olsztyn
  - Travere Investigational Site, Warsaw
  - Travere Investigational Site, Wroclaw
- Portugal (5):
  - Travere Investigational Site, Coimbra
  - Travere Investigational Site, Lisbon
  - Travere Investigational Site, Loures
  - Travere Investigational Site, Setúbal
  - Travere Investigational Site, Vila Nova de Gaia
- South Korea (5):
  - Travere Investigational Site, Seongnam-si, Gyeonggi-do
  - Travere Investigational Site, Anyang-si
  - Travere Investigational Site, Busan
  - Travere Investigational Site, Incheon
  - Travere Investigational Site, Seoul
- Spain (7):
  - Travere Investigational Site, Palma de Mallorca, Balearic Islands
  - Travere Investigational Site, Sagunto, Valencia
  - Travere Investigational Site, Barcelona
  - Travere Investigational Site, Madrid
  - Travere Investigational Site, Seville
  - Travere Investigational Site, Valencia
  - Travere Investigational Site, Zaragoza
- Taiwan (4):
  - Travere Investigational Site, Hualien City
  - Travere Investigational Site, Kaohsiung City
  - Travere Investigational Site, New Taipei City
  - Travere Investigational Site, Taichung
- United Kingdom (18):
  - Travere Investigational Site, Reading, Berkshire
  - Travere Investigational Site, Cambridge, Cambridgeshire
  - Travere Investigational Site, Middlesbrough, Cleveland
  - Travere Investigational Site, Derby, Derbyshire
  - Travere Investigational Site, Brighton, East Sussex
  - Travere Investigational Site, London, Greater London
  - Travere Investigational Site, Manchester, Greater Manchester
  - Travere Investigational Site, Salford, Greater Manchester
  - Travere Investigational Site, Preston, Lancashire
  - Travere Investigational Site, Leicester, Leicestershire
  - Travere Investigational Site, Edinburgh, Scotland
  - Travere Investigational Site, Stoke-on-Trent, Staffordshire
  - Travere Investigational Site, Glasgow, Strathclyde
  - Travere Investigational Site, Carshalton, Surrey
  - Travere Investigational Site, Cardiff, West Glamorgan
  - Travere Investigational Site, Birmingham, West Midlands
  - Travere Investigational Site, Liverpool
  - Travere Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Requests for clinical trial data, including language stating its intended use, should be directed to datarequest@travere.com. If approved, the requested information will be provided to the requestor after signing a data access agreement. Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication. Travere reserves the right to decline or recommend modifications to a request if it does not comply with the data sharing policy or if it is determined that the request is made by a biased source.
Time Frame: Requests can be made following completion of the study and full publication of the study data in a peer reviewed journal for up to 36 months following its publication.
Access Criteria: Requires submission and approval of intended use and a data sharing agreement.

REFERENCES:
- [Derived] Tunnicliffe DJ, Reid S, Craig JC, Samuels JA, Molony DA, Strippoli GF. Non-immunosuppressive treatment for IgA nephropathy. Cochrane Database Syst Rev. 2024 Feb 1;2(2):CD003962. doi: 10.1002/14651858.CD003962.pub3. PMID 38299639
- [Derived] Rovin BH, Barratt J, Heerspink HJL, Alpers CE, Bieler S, Chae DW, Diva UA, Floege J, Gesualdo L, Inrig JK, Kohan DE, Komers R, Kooienga LA, Lafayette R, Maes B, Malecki R, Mercer A, Noronha IL, Oh SW, Peh CA, Praga M, Preciado P, Radhakrishnan J, Rheault MN, Rote WE, Tang SCW, Tesar V, Trachtman H, Trimarchi H, Tumlin JA, Wong MG, Perkovic V; DUPRO steering committee and PROTECT Investigators. Efficacy and safety of sparsentan versus irbesartan in patients with IgA nephropathy (PROTECT): 2-year results from a randomised, active-controlled, phase 3 trial. Lancet. 2023 Dec 2;402(10417):2077-2090. doi: 10.1016/S0140-6736(23)02302-4. Epub 2023 Nov 3. PMID 37931634
- [Derived] Obadina M, Wilson S, Derebail VK, Little J. Emerging Therapies and Advances in Sickle Cell Disease with a Focus on Renal Manifestations. Kidney360. 2023 Jul 1;4(7):997-1005. doi: 10.34067/KID.0000000000000162. Epub 2023 May 31. PMID 37254256
- [Derived] Heerspink HJL, Radhakrishnan J, Alpers CE, Barratt J, Bieler S, Diva U, Inrig J, Komers R, Mercer A, Noronha IL, Rheault MN, Rote W, Rovin B, Trachtman H, Trimarchi H, Wong MG, Perkovic V; PROTECT Investigators. Sparsentan in patients with IgA nephropathy: a prespecified interim analysis from a randomised, double-blind, active-controlled clinical trial. Lancet. 2023 May 13;401(10388):1584-1594. doi: 10.1016/S0140-6736(23)00569-X. Epub 2023 Apr 1. PMID 37015244
- See also: Sponsor Website — http://travere.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The PROTECT study is a 114-week, randomized, multicenter, double-blind (DB), parallel-group, active control study, in participants with Immunoglobulin A nephropathy (IgAN) who had persistent overt proteinuria and remained at high risk of disease progression despite being on a stable dose (or doses) of an Angiotensin converting enzyme inhibitor (ACEI) and/or Angiotensin II receptor blocker (ARB) that was (were) a maximum tolerated dose
Pre-assignment Details: The study was conducted across 3 regions (North America, Europe, and Asia Pacific), 18 countries, and 156 sites. The results presented are based on the double-blind period of the study.
Groups:
- Sparsentan: Participants randomized to Sparsentan received an initial dose of 200 milligrams (mg) (ie, one-half the target dose) tablets over-encapsulated (blinded) with size 00 capsules for the first 2 weeks after randomization. At the Week 2 visit, titration was done up to the target dose (400 mg) based on blood pressure and lack of adverse events (AEs) or after the Week 2 laboratory results were available (ie, between the Week 2 and Week 4 visits).
- Irbesartan: Participants randomized to Irbesartan received an initial dose of 150 mg (ie, one-half the target dose) tablets over-encapsulated (blinded) with size 00 capsules for the first 2 weeks after randomization. At the Week 2 visit, titration was done up to the target dose (300 mg) based on blood pressure and lack of AEs or after the Week 2 laboratory results were available (ie, between the Week 2 and Week 4 visits).
Period: Overall Study
Arm/Group | Sparsentan | Irbesartan
Started | 203 | 203
Received at Least 1 Dose of Study Drug | 202 | 202
Completed (The participant flow presented is based on the double-blind period of the study.) | 199 | 191
Not Completed | 4 | 12
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 4 | 9

BASELINE CHARACTERISTICS:
Population: Full Analysis Set comprised of all participants who were randomized and received at least 1 dose of randomized therapy
Groups:
- Sparsentan: Participants randomized to Sparsentan received an initial dose of 200 mg (ie, one-half the target dose) tablets over-encapsulated (blinded) with size 00 capsules for the first 2 weeks after randomization. At the Week 2 visit, titration was done up to the target dose (400 mg) based on blood pressure and lack of AEs or after the Week 2 laboratory results were available (ie, between the Week 2 and Week 4 visits).
- Total: Total of all reporting groups
Arm/Group | Sparsentan | Irbesartan | Total
Number analyzed (Participants) | 202 | 202 | 404
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.6 (12.76) | 45.4 (12.12) | 46.0 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 59 | 122
  Male | 139 | 143 | 282
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 16 | 33
  Not Hispanic or Latino | 185 | 183 | 368
  Unknown or Not Reported | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 67 | 48 | 115
  Black or African American | 1 | 3 | 4
  White | 130 | 142 | 272
  Other | 4 | 8 | 12
  Multiple | 0 | 1 | 1
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in the Urine Protein/Creatinine (UP/C) at Week 36
Description: 24-hour urine sample was collected for analysis of UP/C via a mixed-model repeated-measures (MMRM) analysis. Missing responses were imputed prior to analysis using multiple imputation. Change from Baseline during the double-blind period in UP/C on the log scale was the dependent variable. Log Baseline UP/C was included as a covariate along with fixed effects for randomized treatment, time (ie, nominal visit in weeks), randomized treatment-by-time interaction, and randomization strata with participants as random effect. Estimates in log scale were back transformed. Baseline was defined as the last non-missing observation on or prior to the start of the dosing. Using Rubin's approach, estimated treatment effects are combined across all imputations to obtain overall estimates.
Time Frame: Baseline (Day 1) and at Week 36
Population: The Primary Analysis Set (PAS) is the subset of the Full Analysis Set at the time of the data extraction for primary analysis. Participants in the PAS were analyzed according to randomized treatment assignment.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Percent change
Groups:
- Sparsentan: Participants randomized to Sparsentan received initial dose of 200 mg (ie, one-half the target dose) tablets over-encapsulated (blinded) with size 00 capsules for the first 2 weeks after randomization. At the Week 2 visit, titration was done up to the target dose (400 mg) based on blood pressure and lack of AEs or after the Week 2 laboratory results were available (ie, between the Week 2 and Week 4 visits).
- Irbesartan: Participants randomized to Irbesartan received initial dose of 150 mg (ie, one-half the target dose) tablets over-encapsulated (blinded) with size 00 capsules for the first 2 weeks after randomization. At the Week 2 visit, titration was done up to the target dose (300 mg) based on blood pressure and lack of AEs or after the Week 2 laboratory results were available (ie, between the Week 2 and Week 4 visits).
Arm/Group | Sparsentan | Irbesartan
Number analyzed (Participants) | 202 | 202
Percent change | -49.77 [-54.98 to -43.95] | -15.05 [-23.72 to -5.39]
Statistical Analysis 1: Comparison: Sparsentan vs Irbesartan; Test type: Other; p < 0.0001, Mixed Models Analysis; Geometric Mean Ratio = 0.59, 95% CI 2-sided [0.51 to 0.69]

2. Secondary Outcome: Total Slope of Estimated Glomerular Filtration Rate (eGFR) Over a 110-week Period
Description: The rate of change in eGFR from Day 1 to Week 110 (ie, over 110 weeks) was analyzed via a mixed-model random coefficients analysis. Missing responses were imputed prior to analysis using multiple imputation. Fixed effects for randomized treatment, Baseline eGFR, time (in weeks), randomized treatment-by-time interaction, and randomization strata were included. In addition, the model also included a random intercept and random slope for each participant. Using Rubin's approach, the estimated treatment effects are combined across all imputations to obtain the overall estimates.
Time Frame: From Day 1 to Week 110
Population: Full Analysis Set.
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliters/minute/1.73square meter/year
Arm/Group | Sparsentan | Irbesartan
Number analyzed (Participants) | 202 | 202
milliliters/minute/1.73square meter/year | -2.9 [-3.58 to -2.24] | -3.9 [-4.59 to -3.13]
Statistical Analysis 1: Comparison: Sparsentan vs Irbesartan; Test type: Other; p = 0.0582, Mixed Models Analysis; Slope difference = 1.0, 95% CI 2-sided [-0.03 to 1.94], Standard Error of Mean 0.50

3. Secondary Outcome: Annualized Slope of eGFR Following the Initial Acute Effect of Randomized Treatment (Chronic Slope)
Description: The rate of change in eGFR from Week 6 to Week 110 (ie, over 104 weeks following the initial acute effect of randomized therapy) was analyzed via a mixed-model random coefficients analysis. Missing responses were imputed prior to analysis using multiple imputation. Fixed effects for randomized treatment, Baseline eGFR, time (in weeks), randomized treatment-by-time interaction, and randomization strata were included. In addition, the model also included a random intercept and random slope for each participant. Using Rubin's approach, the estimated treatment effects are combined across all imputations to obtain the overall estimates.
Time Frame: From Week 6 to Week 110 post randomization
Population: Full Analysis Set.
Measure: Least Squares Mean (95% Confidence Interval); unit: milliliters/minute/1.73square meter/year
Arm/Group | Sparsentan | Irbesartan
Number analyzed (Participants) | 202 | 202
milliliters/minute/1.73square meter/year | -2.7 [-3.43 to -2.05] | -3.8 [-4.60 to -3.07]
Statistical Analysis 1: Comparison: Sparsentan vs Irbesartan; Test type: Other; p = 0.0369, Mixed Models Analysis; Slope difference = 1.1, 95% CI 2-sided [0.07 to 2.12], Standard Error of Mean 0.52

ADVERSE EVENTS:
Time Frame: Up to Week 114
Description: Safety Analysis Set comprised of all participants who were randomized and had received at least 1 dose of randomized therapy. The results presented are based on the double-blind period of the study.
Arm/Group | Sparsentan | Irbesartan
All-Cause Mortality (participants affected / at risk) | 0/202 | 1/202
Serious Adverse Events (participants affected / at risk) | 75/202 | 71/202
Other Adverse Events (participants affected / at risk) | 187/202 | 177/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sparsentan (N=202) | Irbesartan (N=202)
COVID-19 (Infections and infestations) | 42 | 38
Appendicitis (Infections and infestations) | 1 | 2
COVID-19 pneumonia (Infections and infestations) | 1 | 2
Cellulitis (Infections and infestations) | 1 | 2
Cellulitis orbital (Infections and infestations) | 1 | 0
Complicated appendicitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Latent tuberculosis (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Ludwig angina (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 6 | 6
Acute kidney injury (Renal and urinary disorders) | 4 | 1
IgA nephropathy (Renal and urinary disorders) | 1 | 2
Proteinuria (Renal and urinary disorders) | 1 | 2
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1
Perinephric collection (Renal and urinary disorders) | 0 | 1
Prerenal failure (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Radiculopathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal polyp (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 2
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Malaise (General disorders) | 2 | 0
Chest pain (General disorders) | 0 | 1
Hyperplasia (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 1
Target skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Arteriovenous fistula (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Retinal tear (Eye disorders) | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sparsentan (N=202) | Irbesartan (N=202)
COVID-19 (Infections and infestations) | 53 | 46
Upper respiratory tract infection (Infections and infestations) | 18 | 18
Nasopharyngitis (Infections and infestations) | 15 | 16
Urinary tract infection (Infections and infestations) | 7 | 12
Hyperkalaemia (Metabolism and nutrition disorders) | 32 | 26
Gout (Metabolism and nutrition disorders) | 11 | 10
Hyperuricaemia (Metabolism and nutrition disorders) | 7 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 4
Oedema peripheral (General disorders) | 31 | 24
Fatigue (General disorders) | 17 | 11
Diarrhoea (Gastrointestinal disorders) | 10 | 19
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 10 | 8
Nausea (Gastrointestinal disorders) | 10 | 5
Blood creatine phosphokinase increased (Investigations) | 15 | 10
Blood creatinine increased (Investigations) | 10 | 14
Lipase increased (Investigations) | 12 | 9
Alanine aminotransferase increased (Investigations) | 10 | 8
Headache (Nervous system disorders) | 27 | 26
Dizziness (Nervous system disorders) | 30 | 13
Proteinuria (Renal and urinary disorders) | 13 | 15
Renal impairment (Renal and urinary disorders) | 7 | 12
Acute kidney injury (Renal and urinary disorders) | 12 | 5
Hypertension (Vascular disorders) | 22 | 28
Hypotension (Vascular disorders) | 26 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 8
Anaemia (Blood and lymphatic system disorders) | 16 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT03762850/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/50/NCT03762850/SAP_001.pdf